CLINICAL TRIAL: NCT06298045
Title: Effectiveness and Impact on Quality of Life of a Combination of Trimetazidine With One Hemodynamic Agent (ß-blocker or Ca-channel Blocker), in Patients Recently Diagnosed With Stable Angina and Still Symptomatic Despite First Line Hemodynamic Therapy: a Prospective, International, Non-interventional Study.
Brief Title: Effectiveness of a Combination of Trimetazidine With One Hemodynamic Agent in Patients Recently Diagnosed With Stable Angina and Still Symptomatic Despite First Line Hemodynamic Therapy
Status: Recruiting | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-06790-002
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stable Angina
Keywords: Symptomatic Stable Angina; Adherence; prospective, international, non-interventional study; Quality of life
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess in recently diagnosed stable Angina patients symptomatic despite first line hemodynamic therapy, the effect of a combination of this hemodynamic agent with a metabolic one (trimetazidine). The treatment effect will be measured by the reduction of patients' angina symptoms, physical limitation and an improvement of quality of life using the Seattle Angina Questionnaire-7 items (SAQ-7) Patients will be also proposed to complete a BEAMER (BEhavioral and Adherence Model for improving quality, health outcomes and cost-Effectiveness of healthcaRe) questionnaire which will contribute to a separate research project developed by the Innovative Medicines Initiative (IMI). Analysis of the BEAMER questionnaires will be performed outside the study by the IMI BEAMER Consortium for BEAMER purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Male and female recently diagnosed symptomatic stable Angina patients
* Age ≥18 years old
* Patient already treated by one first line antianginal haemodynamic agent (ß-blocker or Ca-channel blocker) (according to CCS management guidelines 2019) and still symptomatic after initiation of this antianginal treatment.
* Patient for whom the physician intends to prescribe trimetazidine based on her/his daily medical practice in the management of symptomatic Angina pectoris, respecting the SmPC in force in the country. Such treatment decision must be taken independently from the participation of the patient in the study.
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Any contra-indication to trimetazidine according to SmPC
* Patient already treated with trimetazidine before entry into the study.
* Pregnancy or intention to become pregnant or lactating women during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female recently diagnosed symptomatic stable Angina patients.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of angina symptoms via the summary score of SAQ-7 | from 2 weeks to 4 months

SECONDARY OUTCOMES:
CCS angina grading post-inclusion | from 2 weeks to 4 months
Tolerance ( Adverse Events) | from 2 weeks to 4 months
  Number of patients with adverse events
Tolerance ( Serious Adverse Events) | from 2 weeks to 4 months
  Number of patients with serious adverse events
Adherence to the antianginal treatment combination under evaluation | from 2 weeks to 4 months
  Adherence is measured by MARS-5 (a continuous variable)

CONTACTS AND LOCATIONS:
Locations (1):
- Thera Card Srl, Brasov, Romania